CLINICAL TRIAL: NCT06220682
Title: Role of Endothelial Nitric Oxide Synthase Polymorphic Gene (c.894 G>T) in Coronary Artery Dilation Disease
Brief Title: Endothelial NO Synthase Polymorphic Gene in Coronary Artery Dilation Disease
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Farouk, Lecturer of critical care, Cairo University
Other Study IDs: Kasralainy school of medicine
Record Dates: First submitted 2023-12-27; First posted 2024-01-24 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Ectasia
MeSH Terms: conditions — Coronary Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- normal group: 25 patients angiographically normal coronaries
  Interventions: Diagnostic Test: The specific genetic PCR laboratory test were performed for all selected patients for eNOS SNPs
- atherosclerotic non dilated group: 25 patients angiographically had atherosclerotic plaques with no coronary dilatations
- dilated non atherosclerotic group: 25 patients angiographically involved coronary dilatations with no atherosclerotic plaques
- dilated atherosclerotic group: 25 patients angiographically had both coronary dilatations and atherosclerotic plaques
  Interventions: Diagnostic Test: The specific genetic PCR laboratory test were performed for all selected patients for eNOS SNPs

INTERVENTIONS:
Diagnostic Test: The specific genetic PCR laboratory test were performed for all selected patients for eNOS SNPs — using Real-Time PCR (QuantStudioTM 3 Real-Time PCR) with an allele-specific fluorogenic oligonucleotide probe and a TaqMan pre-designed SNP Genotyping assay
  Groups: dilated atherosclerotic group; normal group

SUMMARY:
Introduction: The coronary artery dilatations disease (Coronary artery aneurysm/coronary artery ectasia) characterized by inappropriate coronary artery dilations. (c.894G>T) is a gene polymorphism that may decreases eNOS enzyme activity which increases the risk for coronary heart disease by affecting released (NO) molecules. One of the most researched variations in eNOS gene is c.894G>T polymorphism, which changes amino acid sequence at position 298 from Glu (GAG) to Asp (GAT), nevertheless, its role in Coronary dilatations disease still uncertain.

Aim of study: To study correlation between the c.894G>T gene polymorphism and angiographically dilated coronary artery (CAA/CAE), as well as to determine whether there is any association between this polymorphism and atherosclerotic CAD.

Methodology: A comparative study on 100 patients with acute coronary syndrome who underwent coronary angiography from December 2020 to June 2022. According to standard angiographic views and expert opinions, patients were divided as, 25 patients normal, 25 patients had only atherosclerotic coronary artery disease, 25 patients had dilated coronaries (CAA/CAE) without atherosclerosis and 25 patients had dilated coronaries with atherosclerotic coronary artery disease. The specific genetic PCR laboratory test were performed for eNOS SNPs (single nucleotide polymorphism) namely, 894G > T (Glu298Asp; rs 1799983), using Real-Time PCR.

DETAILED DESCRIPTION:
Aim of Work We aim at determining the potential correlations between polymorphism of nitric oxide gene (c.894G>T) and angiographically dilated coronary arteries (coronary artery aneurysm or ectasia), as well as to determine if there is any link to atherosclerotic coronary diseases (ACAD).

Methodology:

Based on standard coronary angiographic views, two experienced independent operators evaluated the presence of coronary artery dilatations (CAA, CAE) and associated atherosclerotic CAD in all patients' angiograms.

Inclusion criteria Patients who have angiographically coronary artery dilatations (coronary artery aneurysm or ectasia) (CAA/CAE) with or without angiographic evidence of atherosclerotic CAD.

Another group of patients with angiographically normal or atherosclerotic coronaries without evidence of dilatation.

Exclusion criteria Patients with secondary coronary dilatations after balloon angioplasty, coronary stent implantation, patients with coronary artery bypass surgery who have post CABG native coronary dilatations, all were excluded from this study.

Definitions CAE refers to a diffuse dilatation affecting more than 1/3 of length of CA where its diameter is 1.5 greater than subsequent healthy coronary portion [1, 2, 3].

CAA is less common clinical finding that is described as dilation at the CAs that is < 1/3 of the length of the CA also with diameter 1.5 greater than normal length of nearby part [1, 2, 3, 4].

Laboratory method and genetic analysis The specific genetic PCR laboratory test were performed for all selected patients for eNOS SNPs (single nucleotide polymorphism) namely, 894G > T (Glu298Asp; rs 1799983), using Real-Time PCR (QuantStudioTM 3 Real-Time PCR) with an allele-specific fluorogenic oligonucleotide probe and a TaqMan pre-designed SNP Genotyping assay (TaqMan technique; Applied Biosystems, Germany), The fluorogenic dyes employed to achieve allelic discrimination were FAM (6-carboxy-fluorescein) and VIC (Applied Biosystems proprietary dye). a total reaction volume of 25 L (12.5L TaqMan® Genotyping Master Mix) (2x) - 1.25 µL TaqMan genotyping assay(20x) -5.0µL genomic DNA- 6.25µL DNase-free, RNasefree water) is used to perform PCR.

Primary outcome: To study correlation between the c.894G>T gene polymorphism and angiographically dilated coronary artery (CAA/CAE) Secondary outcome: To determine whether there is any association between this polymorphism and atherosclerotic CAD.

Statistical analysis SPSS v.21 statistical package was used to code and entering data, where it described as number and percent for qualitative mean and standard deviation (SD) for normally distributed data while median and inter quintile rang (IQR) chosen for non-normally distributed quantitative data.

Comparisons for qualitative variables between groups was mad by chi-square or fissure exact tests, while comparisons across normally distributed quantitative variables were done using analysis of variance and post hock 2khs test, and quantitative variables which is not normally distributed, where compared using (non-parametrical croscal wise and Mann-Whitney u tests), statistically significant considered when P. values was below or equal (0.05).

ELIGIBILITY:
Inclusion Criteria:

Patients who have angiographically coronary artery dilatations (coronary artery aneurysm or ectasia) (CAA/CAE) with or without angiographic evidence of atherosclerotic CAD.

Another group of patients with angiographically normal or atherosclerotic coronaries without evidence of dilatation.

Exclusion Criteria:

Patients with secondary coronary dilatations after balloon angioplasty, coronary stent implantation, patients with coronary artery bypass surgery who have post CABG native coronary dilatations, all were excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The total populations in our study were 100 patients, divided into 4 groups depends on angiographic results:
  Group (1): 25 patients angiographically normal coronaries (normal group). Group (2): 25 patients angiographically had atherosclerotic plaques with no coronary dilatations (atherosclerotic non dilated group).
  Group (3): 25 patients angiographically involved coronary dilatations with no atherosclerotic plaques (dilated non atherosclerotic group).
  Group (4): 25 patients angiographically had both coronary dilatations and atherosclerotic plaques (dilated atherosclerotic group).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
: To study correlation between the c.894G>T gene polymorphism and angiographically dilated coronary artery (CAA/CAE) | 1 year
  : To study correlation between the c.894G>T gene polymorphism and angiographically dilated coronary artery (CAA/CAE)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mowafy, MD, Study Chair — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No